CLINICAL TRIAL: NCT02496078
Title: A Phase 3 Evaluation of Daclatasvir and Asunaprevir in Treatment-naive Subjects With Chronic Hepatitis C Genotype 1b Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI447-114
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active dual arm (Active Comparator): Daclatasvir in tablet form at the dose of 60 mg QD and Asunaprevir in soft capsule form at the dose of 100 mg BID from day 1 to 12 week
  Daclatasvir in tablet form at the dose of 60 mg QD and Asunaprevir in soft capsule form at the dose of 100 mg BID from 12 to 24 week and follow up to week 48
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir
- Placebo arm (Placebo Comparator): Daclatasvir placebo in tablet form QD and Asunaprevir placebo in soft capsule form BID from day 1 to 12 week
  Daclatasvir in tablet form at the dose of 60 mg QD and Asunaprevir in soft capsule form at the dose of 100 mg BID from 12 to 36 week and follow up to week 60
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir

INTERVENTIONS:
Drug: Daclatasvir — Daclatasvir tablet 60mg
Drug: Asunaprevir — Asunaprevir soft capsule 100 mg

SUMMARY:
The purpose of this study is to determine whether a regimen consisting of daclatasvir and asunaprevir is effective in treatment-naive patients with chronic hepatitis genotype 1b infection.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients chronically infected with HCV Genotype 1b
* No previous exposure to any interferon formulation, Ribavirin (RBV), and HCV direct acting antiviral agent
* HCV RNA viral load ≥ 10,000 IU/mL at screening
* Seronegative for HIV and HBsAg
* BMI of 18-35 kg/m2, inclusive
* Patients with compensated cirrhosis are permitted

Exclusion Criteria:

* Infection with HCV other than genotype (GT) -1b
* Evidence of decompensated liver disease including, but not limited to, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
* Evidence of a medical condition contributing to chronic liver disease other than HCV
* Diagnosed or suspected hepatocellular carcinoma or other malignancies
* Uncontrolled diabetes or hypertension
* History of moderate to severe depression. Well-controlled mild depression is allowed
* Confirmed alanine aminotransferase (ALT) ≥ 5x Upper Limit of Normal (ULN)
* Confirmed platelet count < 50,000 cells/mm3
* Confirmed hemoglobin < 8.5 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of treated subjects randomized to Active Dual therapy with Sustained Virologic Response (SVR12) | Post-treatment Week 12
  HCV RNA < Lower limit of quantitation (LLOQ) target detected (TD) or target not detected (TND) at follow-up Week 12

SECONDARY OUTCOMES:
Proportion of subjects with anemia on active Dual therapy | Post-treatment Week 12
Proportion of subjects with neutropenia on active Dual therapy | Post-treatment Week 12
Proportion of subjects with thrombocytopenia on active Dual therapy | Post-treatment Week 12
On treatment safety, as measured by frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Post-treatment week 12
Differences in rates of selected Grade 3-4 laboratory abnormalities for hematology between treatments (DCV + Asunaprevir (ASV) vs PBO) | first 12 weeks on treatment
Differences in rates of selected Grade 3-4 laboratory abnormalities for liver function between treatments (DCV + Asunaprevir (ASV) vs PBO) | first 12 weeks on treatment
Proportion of subjects with SVR12 by the rs12979860 single nucleotide polymorphism (SNP) in the interleukin (IL) -28B gene for each cohort | Post-treatment visit week 12
Proportion of subjects with hepatitis C virus (HCV) RNA < LLOQ-TD/TND in each arm at various intervals after the initiation of active Dual therapy | post-treatment visit Week 24
Proportion of subjects who achieve HCV RNA < LLOQ-TND at each arm at various intervals after the initiation of active Dual therapy | post-treatment visit Week 24
Proportion of treated subjects with SVR12 for subjects randomized to placebo | Post-treatment visit week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- China (13):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Shijiazhuang, Hebei
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Zhenjiang, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Qingdao, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Xi’an, Shanxi
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Beijing
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- South Korea (2):
  - Local Institution, Busan
  - Local Institution, Seoul

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx